CLINICAL TRIAL: NCT04968769
Title: Comparison of Ischemic Compression Therapy and Kinesiotaping on Blood Flow, Tissue Stiffness, Pain and Range of Motion in Chronic Neck Pain
Brief Title: Comparison of Ischemic Compression Therapy and Kinesiotaping in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 21/19
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Neck Pain
Keywords: Trapezius muscle; trigger point; ultrasonographic imaging; blood flow; chronic pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Acupressure; Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ischemic compression and exercise (Experimental): Individuals were positioned in a comfortable position in a chair with back support. By palpating the UT muscle, first the taut band and then the active TP on the muscle were determined. Before starting the treatment, , a statement was made to the individual that "you will soon feel a high level of pain with pressure, and at the same time, you may feel pain, tingling, pricking in additional areas (head-neck-shoulder-arm), after a while the pain will decrease and disappear. In this process, try to stay as steady as possible and breathe regularly and calmly.'' The highest level of pressure that the patient could tolerate was applied to the determined TP with the thumb. Pressure time will be in the range of at least 10-20 seconds and at most 60 seconds; It was terminated after the therapist felt complete relaxation in the tissue under his thumb or after the patient received the return of "pain completely disappeared"
  Interventions: Other: ischemic compression; Other: exercise
- kinesio taping and exercise (Experimental): While performing KT, the individual was seated in a comfortable and upright position in a chair with back support. The subject was asked to bring his hand to his back in internal rotation of the shoulder of the taped side and to bring his head to the contralateral lateral flexion and contralateral rotation so that the UT muscle was in a tense position. KT was applied using 'muscle inhibition technique' to ensure correct contraction of the muscle with muscle length/tension optimization, to target the reduction of excessive muscle tension, and to increase circulation with the effects of the tape on the skin. In this technique, to inhibit the muscle, the tape direction is from the muscle insertion to the origin. KT was performed 5 cm below the acromion to the protuberantia occipitalis with 10% tension
  Interventions: Other: kinesio taping; Other: exercise
- exercise (Active Comparator): In order for all the exercises to be done correctly and not to cause any pain, the individuals were asked to perform the movements in front of the mirror. Posture exercises given the individuals for scapular retraction. During the posture exercises individual was positioned in a chair without back support. By counting 5 it was requested to do 10 repetitions of each exercise. For the UT muscle stretching, individuals were asked to hold their right ear with their left hand over their head while sitting on a back-supported chair with their hips and back fully resting on the chair, and to bring their left ear closer to their left shoulder with the help of their hand and count to 20 from the outside.
  Interventions: Other: exercise

INTERVENTIONS:
Other: ischemic compression — manual therapy
  Arms: ischemic compression and exercise
Other: kinesio taping — elastic therapeutic taping
  Arms: kinesio taping and exercise
Other: exercise — posture exercises

SUMMARY:
Objective: The purpose of this study was to compare the effects of ischemic compression (IC) and kinesio taping (KT) treatments on blood flow, tissue stiffness and thickness, pain, and joint range of motion on the upper trapezius muscle of individuals with chronic neck pain.

Methods: In this study 22 individuals between the ages of 20-35 were randomly assigned to 3 groups: Group1, which received IC; Group2, received KT; Group3 (control) received exercise, for 2 days and 4 weeks. Pain was measured with VAS, pain threshold with J-Tech Algometer, range of motion with BASELINE Digital Inclinometer, ultrasonographic measurements for blood flow, tissue stiffness and tissue thickness using Acuson S3000. All measurements were performed twice; before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* A score ar least 3 and above 3 on the Visual analogue scale
* Presence of palpable taut band and at least one trigger point on the taut band
* Presence of referred pain with palpation of the trigger point

Exclusion Criteria:

* Analgesic use within the previous 24hours
* History of cervical surgery
* Receiving myofascial pain treatment within the previous month of the study

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
pain intensity | 4 weeks
  Visual Analogue Scale: Individuals were asked to mark the intensity of neck pain on the scale, defining the visual analog scale as 0 "absence of pain-no pain" and 10 "unbearable-worst pain". The distance between the sign of the individual and the 0 point was measured and recorded
pain threshold | 4 weeks
  Individuals were asked to sit in a comfortable position in a chair with back support. Before starting the measurement, a statement was made to the individual that "when the pressure sensation turns into pain, give a stop warning". The measurement was repeated 3 times and the average value was recorded. A 30-second interval was taken between measurements to prevent temporal summation. Measurements were taken over the UT muscle of the dominant extremity with the J-TECH USA Commander Algometer device
range of motion | 4 weeks
  For ROM measurements individuals were asked to sit on a chair with back support with hands on thighs, shoulders free, hips and knees 90 flexed. For neck flexion and extension movements, the inclinometer was placed on the head of the individual in the sagittal plane, and for the right and left lateral flexion movements, the inclinometer was placed in the frontal plane. For neck rotation measurements, the individual was placed in a supine and relaxed position. The inclinometer was placed on the forehead of the head in the transverse plane. For each measurement, the individual was asked to actively perform the movement to be measured, and the average value was recorded for each parameter by repeating it 3 times. Before each measurement, the inclinometer was restarted after it was positioned over the individual's head. Measurements were made with the BASELİNE Digital Inclinometer device
Ultrasonographic Measurements | 4 weeks
  Ultrasonographic measurements Using a 9L4 MHz (Megahertz) linear transducer (Acuson S2000, Siemens Healthcare, Erlangen, Germany) with sufficient amount of gel, the upper fibers of the dominant tar
  trapezius muscle were aligned longitudinally to the muscle fibers inside the transducer UT muscle with a dorsal approach at the mid-clavicular line level. The thickness of the UT muscle, B mode, peak systolic velocity (PV-cm/s) data from the transverse cervical artery, color Doppler ultrasound (RDUS) and the UT muscle fibers of the muscle again in quantitative ARFI mode (Virtual Touch Quantification®, VTq) for tissue stiffness assessment. Mean VTq values were calculated by taking VTq (m/sec) measurements 10 times.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided